CLINICAL TRIAL: NCT05554796
Title: Endoscopic Stapedotomy: Classic Versus Reversal Technique
Brief Title: Endoscopic Classic Versus Reversal Stapedotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Hemdan, Lecturer of Otorhinolaryngology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.21.11.1758
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Otosclerosis of Middle Ear

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic classic stapedotomy (Experimental): This groups contains 30 patients and will undergo classic stapedotomy
  Interventions: Procedure: Endoscopic classic stapedotomy
- Endoscopic reversal stapedotomy (Experimental): This groups contains 30 patients and will undergo reversal stapedotomy
  Interventions: Procedure: Endoscopic reversal stapedotomy

INTERVENTIONS:
Procedure: Endoscopic classic stapedotomy — Patients in this group will undergo classic stapedotomy starting with removal of stapes superstructure then perforation of footplate and finally insertion of the Teflon piston.
  Arms: Endoscopic classic stapedotomy
Procedure: Endoscopic reversal stapedotomy — Patients in this group will undergo reversal stapedotomy where perforation of footplate and insertion of Teflon piston will be done at the beginning followed by removal of stapes superstructure.
  Arms: Endoscopic reversal stapedotomy

SUMMARY:
Aim of The Work The aim of this study is to compare hearing outcome and surgical complications between classic and reversal endoscopic stapedotomy.

Patients and Methods

Study design:

This study is a randomized clinical study and will be carried out at Otorhinolaryngology department at Mansoura University Hospitals. The study will be conducted among 60 patients with otosclerosis who will undergo endoscopic stapedotomy. The patients will be divided into two groups. The first group (group 1) 30 patients will undergo endoscopic classic stapedotomy while the second group (group 2) 30 patients will undergo endoscopic reversal stapedotomy.

The two groups will compared to each other as regard, A. Intra-operative time (in minutes) B. Hearing outcome. C. Surgical complications

DETAILED DESCRIPTION:
Aim of The Work The aim of this study is to compare hearing outcome and surgical complications between classic and reversal endoscopic stapedotomy.

Patients and Methods

Study design:

This study is a randomized clinical study and will be carried out at Otorhinolaryngology department at Mansoura University Hospitals. The study will be conducted among 60 patients with otosclerosis who will undergo endoscopic stapedotomy. The patients will be divided into two groups. The first group (group 1) 30 patients will undergo endoscopic classic stapedotomy while the second group (group 2) 30 patients will undergo endoscopic reversal stapedotomy.

Inclusion criteria:

Patients with history of gradual progressive hearing loss with normal otoscopy. No history of ear discharge. No history of ipsilateral ear surgery. Air bone gap >20 dB with lost stapedial reflex

Exclusion criteria:

Cases who did not meet the inclusion criteria. Revision cases. Cases that lost to follow up. All cases with narrow oval window niche or obliterated footplate, because those are the contraindications of reversal technique as described by Fisch (Fisch et al., 1994).

The two groups will compared to each other as regard,

A. Intra-operative time (in minutes):

Starting from the incision till repositioning of the flap. B. Hearing outcome. Hearing outcomes will include the average air conduction pure-tone threshold (in dB HL) and a word recognition score (WRS, in %). The data will be reported on a scattergram relating average air conduction pure-tone threshold to the WRS.

Preoperative and postoperative air conduction (AC) and bone conduction (BC) thresholds will be recorded at frequencies of 0.5, 1, 2, and 3 khz. The air-bone gap (ABG) will be recorded as the difference between AC and BC thresholds. Postoperative air bone gap will be graded as grade A (0-10 dB), grade B (11-20 dB), grade C (21-30 dB) and grade D (>30 dB).

C. Surgical complications:

Vertigo. Incus subluxation. Corda tympani nerve injury. Tympanic membrane tear. Perilymph gusher. Floating footplate. Postoperative pain. Perilymph fistula. Immediate or late sensory neural hearing loss.

Method:

All cases planned to be included in this study will be subjected to:

History taking:

Personal history, past history of medical diseases, past history of surgery and family history.

Examination: routine ENT examination to exclude any other ear disease.

Investigations:

A. PTA ,Tympanogram. B. Lab investigations: Pre-operative full lab(CBC, INR, LFT,virology)

Surgeries:

Patients will be operated under local anesthesia, and the transcanal approach will be the standard approach in both groups. Zero and thirty degree, 4 mm diameter, 18 cm length endoscopes and camera will be used.

Group 1:

Patients in this group will undergo classic stapedotomy where removal of stapes superstructure will be performed in the beginning followed by perforation of footplate and finally insertion of the Teflon piston.

Group 2:

Patients in this group will undergo reversal stapedotomy where perforation of footplate and insertion of Teflon piston will be done at the beginning followed by removal of stapes superstructure.

Statistical analysis:- Data analysis will be carried out using statistical software program (SPSS for Windows, version 28, USA). Variables will be presented as mean ± standard deviations (SDs), and percentages. The preoperative and postoperative hearing results (AC and BC and ABG) will be compared utilizing the paired t-test. Statistical significance will be considered at P <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of gradual progressive hearing loss with normal otoscopy.
* No history of ear discharge.
* No history of ipsilateral ear surgery.
* Air bone gap >20 dB with lost stapedial reflex

Exclusion Criteria:

* Cases who did not meet the inclusion criteria.
* Revision cases.
* Cases that lost to follow up.
* All cases with narrow oval window niche or obliterated footplate, because those are the contraindications of reversal technique as described by Fisch (Fisch et al., 1994).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Average air conduction pure-tone threshold | 3 months
  The average air conduction pure-tone threshold (in dB HL) will be calculated from pure-tone audiometry and presented in decibels (dB)
Word recognition score | 3 months
  The word recognition score will be calculated from the the speech audiometry and presented as percentage (%)
Average air bone gap | 3 months
  Preoperative and postoperative air conduction (AC) and bone conduction (BC) thresholds will be recorded at frequencies of 0.5, 1, 2, and 3 khz. The air-bone gap (ABG) will be recorded as the difference between AC and BC thresholds. Postoperative air bone gap will be graded as grade A (0-10 dB), grade B (11-20 dB), grade C (21-30 dB) and grade D (>30 dB).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hemdan, MD, Principal Investigator — Lecturer of Otorhinolaryngology
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt